CLINICAL TRIAL: NCT02877433
Title: Clinical Performance of 4 mm Short Distal Implants in Fixed Cross-Arch Prostheses - An Open, Randomized, Controlled Study
Brief Title: 4 mm Implants in Fixed Cross-Arch Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR 03/15
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2024-07

CONDITIONS: Jaw Edentulous
Keywords: Small diameter implant; Cross-arch prostheses
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roxolid short implant, 4 mm length (4) (Active Comparator): Straumann Tissue Level Ø4.1 mm RN SLActive Roxolid Standard Plus Implants available in lengths 4mm, 10mm, 12mm and 14mm
  Interventions: Device: Roxolid short implant, 4 mm length (4)
- Roxolid short implant, 4 mm length (2) (Experimental): Straumann Tissue Level Ø4.1 mm RN SLActive Roxolid Standard Plus Implants available in lengths 4mm, 10mm, 12mm and 14mm
  Interventions: Device: Roxolid short implant, 4 mm length (2)

INTERVENTIONS:
Device: Roxolid short implant, 4 mm length (4) — Placement of a combination of four short implants (in positions 35/45, 36/46) as distal support and two implants of conventional length (in positions 33/43) in the interforaminal region, in order to support a cross-arch fixed screw-retained prosthesis.
  Arms: Roxolid short implant, 4 mm length (4)
Device: Roxolid short implant, 4 mm length (2) — Placement of a combination of two short implants (in positions 36/46) as distal support and two implants of conventional length (in positions 33/43) in the interforaminal region, in order to support a cross-arch fixed screw-retained prosthesis.
  Arms: Roxolid short implant, 4 mm length (2)

SUMMARY:
This study aims to compare the clinical performance of 4 mm short implants supporting cross-arch fixed reconstructions in the edentulous mandible either with a combination of two short implants as distal support and two implants of conventional length placed in the interforaminal region, or with a combination of four short implants as distal support and two interforaminal implants of conventional length.

DETAILED DESCRIPTION:
This is a post-market, multi-center, prospective, open, randomized controlled clinical study. The total study duration for each patient should be 36 ± 2 months.

Roxolid Standard Plus Implants, 4 mm, Ø 4.1 mm, SLActive will be placed in positions 36/46 or 35/45, 36/46.

Roxolid Standard Plus Implants, Ø 4.1 mm, SLActive, in lengths of 10, 12 and 14 mm will be placed in positions 33/43.

In total 10 visits per patient are scheduled in this study. Implant survival, implant success, prosthetic survival and success, and adverse events (AEs) will be assessed.

All products are CE-(Conformité Européenne, meaning European Conformity) marked and used within its intended use.

Two centers in Switzerland and Northern Ireland will participate. The study and any amendments will be performed according to International Organization for Standardization (ISO) 14155:2011, local legal and regulatory requirements and conform to the Declaration of Helsinki (last revision Fortaleza 2013)

ELIGIBILITY:
Inclusion Criteria:

* Males and females with at least 18 years of age (including 18 years)
* Subject must have voluntarily signed the informed consent, are willing and able to attend scheduled follow-up visits, and agree that the encoded data will be collected and analyzed
* Fully edentulous (latest extraction in the mandible should be performed at least 12 weeks before implant placement) that can be restored with a complete denture
* Atrophic jaw bone in the posterior area, sufficient bone height and width to permit insertion of four short implants, 4 mm in regions of the first molar and second premolar on both sides and two standard length implants in the canine region

Exclusion Criteria:

* Patients with inadequate bone volume and/or quality
* Uncontrolled systemic disease that would interfere with dental implant therapy (e.g. uncontrolled diabetes)
* Any contraindications for oral surgical procedures
* History of local irradiation therapy in the head / neck area
* Patients who smoke >10 cigarettes per day or tobacco equivalents, chew tobacco or have ≥ 20 pack years
* Medical conditions requiring chronic high dose steroid therapy or high dose anti-resorptive treatment
* Subjects who have undergone administration of any investigational device within 30 days of enrollment in the study
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Cognitive impairment that would interfere with the ability to perform adequate oral hygiene (assessed by the Ottawa 3DY scale)
* Patients with chronic pain
* Patients with HIV and/ or Hepatitis infection
* Severe bruxing or clenching habits
* Patients with inadequate oral hygiene or unmotivated for adequate home care (Denture Plaque Index (DPI) ≥ 5)
* Patients with drug or alcohol abuse
* Patients with allergies or hypersensitivity to chemical ingredients of titanium-zirconium alloy
* Major simultaneous augmentation procedures. Dehiscence of a vertical distance of more than 3 mm
* A woman who is pregnant or planning to become pregnant at any point during the study duration

Secondary Exclusion Criteria:

* Patients with inadequate bone volume and/or quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Implant survival | 12 months after baseline
  A surviving implant is defined as an implant in place at the time of the follow-up. Any implant loss shall be assessed as an early loss (implant fails before being osseointegrated) or late loss (after being osseointegrated)

SECONDARY OUTCOMES:
Implant success will be evaluated according to Buser | 12 and 36 months after baseline
  A particular implant will be considered successful if all of the following success criteria according to Buser et al. (Buser et al. 1991) apply:
  * Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (painful sensation)
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics)
  * Absence of implant mobility on manual palpation
  * Absence of any continuous peri-implant radiolucency
Prosthetic survival & success | 12 and 36 months after baseline
  During the prosthodontic examination, the implant supported prostheses will be examined for any complications and failures as adapted from the ITI Treatment Guide Volume 8 (Brägger & Heitz-Mayfield 2015)
Crestal bone level change at the implant site (mesial and distal) | 12 and 36 months after baseline
  Mesial and distal implant bone levels will be evaluated on a panoramic radiograph at baseline, 12 and 36 months after implant loading

OTHER OUTCOMES:
Implant survival | 36 months after baseline
  A surviving implant is defined as an implant in place at the time of the follow-up. Any implant loss shall be assessed as an early loss (implant fails before being osseointegrated) or late loss (after being osseointegrated)

CONTACTS AND LOCATIONS:
Overall Officials: Julia-Gabriela Wittneben, Dr., Principal Investigator — University of Bern, Department of Reconstructive Dentistry and Gerodontology
Locations (2):
- University of Bern, Department of Reconstructive Dentistry and Gerodontology, Bern, Switzerland
- Queens University Belfast, School of Medecine, Dentistry and Biomedical Sciences, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrektsson T, Zarb GA. Current interpretations of the osseointegrated response: clinical significance. Int J Prosthodont. 1993 Mar-Apr;6(2):95-105. PMID 8329101
- [Background] Allen F, Locker D. A modified short version of the oral health impact profile for assessing health-related quality of life in edentulous adults. Int J Prosthodont. 2002 Sep-Oct;15(5):446-50. PMID 12375458
- [Background] Ambjornsen E, Valderhaug J, Norheim PW, Floystrand F. Assessment of an additive index for plaque accumulation on complete maxillary dentures. Acta Odontol Scand. 1982;40(4):203-8. doi: 10.3109/00016358209019813. PMID 6958165
- [Background] Annibali S, Cristalli MP, Dell'Aquila D, Bignozzi I, La Monaca G, Pilloni A. Short dental implants: a systematic review. J Dent Res. 2012 Jan;91(1):25-32. doi: 10.1177/0022034511425675. Epub 2011 Oct 27. PMID 22034499
- [Background] Benzing U, Weber H, Simonis A, Engel E. Changes in chewing patterns after implantation in the edentulous mandible. Int J Oral Maxillofac Implants. 1994 Mar-Apr;9(2):207-13. PMID 8206557
- [Background] Brennan M, Houston F, O'Sullivan M, O'Connell B. Patient satisfaction and oral health-related quality of life outcomes of implant overdentures and fixed complete dentures. Int J Oral Maxillofac Implants. 2010 Jul-Aug;25(4):791-800. PMID 20657876
- [Background] Buser D, Weber HP, Bragger U, Balsiger C. Tissue integration of one-stage ITI implants: 3-year results of a longitudinal study with Hollow-Cylinder and Hollow-Screw implants. Int J Oral Maxillofac Implants. 1991 Winter;6(4):405-12. PMID 1820309
- [Background] Carlsson GE, Lindquist LW. Ten-year longitudinal study of masticatory function in edentulous patients treated with fixed complete dentures on osseointegrated implants. Int J Prosthodont. 1994 Sep-Oct;7(5):448-53. PMID 7802913
- [Background] de Grandmont P, Feine JS, Tache R, Boudrias P, Donohue WB, Tanguay R, Lund JP. Within-subject comparisons of implant-supported mandibular prostheses: psychometric evaluation. J Dent Res. 1994 May;73(5):1096-104. doi: 10.1177/00220345940730051201. PMID 8006237
- [Background] Hamdan NM, Gray-Donald K, Awad MA, Johnson-Down L, Wollin S, Feine JS. Do implant overdentures improve dietary intake? A randomized clinical trial. J Dent Res. 2013 Dec;92(12 Suppl):146S-53S. doi: 10.1177/0022034513504948. Epub 2013 Oct 24. PMID 24158335
- [Background] Heydecke G, Locker D, Awad MA, Lund JP, Feine JS. Oral and general health-related quality of life with conventional and implant dentures. Community Dent Oral Epidemiol. 2003 Jun;31(3):161-8. doi: 10.1034/j.1600-0528.2003.00029.x. PMID 12752541
- [Background] Ikebe K, Matsuda K, Morii K, Furuya-Yoshinaka M, Nokubi T, Renner RP. Association of masticatory performance with age, posterior occlusal contacts, occlusal force, and salivary flow in older adults. Int J Prosthodont. 2006 Sep-Oct;19(5):475-81. PMID 17323726
- [Background] John MT, Patrick DL, Slade GD. The German version of the Oral Health Impact Profile--translation and psychometric properties. Eur J Oral Sci. 2002 Dec;110(6):425-33. doi: 10.1034/j.1600-0722.2002.21363.x. PMID 12507215
- [Background] Millwood J, Heath MR. Food choice by older people: the use of semi-structured interviews with open and closed questions. Gerodontology. 2000 Jul;17(1):25-32. doi: 10.1111/j.1741-2358.2000.00025.x. PMID 11203509
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Muller F, Duvernay E, Loup A, Vazquez L, Herrmann FR, Schimmel M. Implant-supported mandibular overdentures in very old adults: a randomized controlled trial. J Dent Res. 2013 Dec;92(12 Suppl):154S-60S. doi: 10.1177/0022034513509630. Epub 2013 Oct 24. PMID 24158342
- [Background] Muller F, Hernandez M, Grutter L, Aracil-Kessler L, Weingart D, Schimmel M. Masseter muscle thickness, chewing efficiency and bite force in edentulous patients with fixed and removable implant-supported prostheses: a cross-sectional multicenter study. Clin Oral Implants Res. 2012 Feb;23(2):144-150. doi: 10.1111/j.1600-0501.2011.02213.x. Epub 2011 Jun 2. PMID 21631592
- [Background] Rashid F, Awad MA, Thomason JM, Piovano A, Spielberg GP, Scilingo E, Mojon P, Muller F, Spielberg M, Heydecke G, Stoker G, Wismeijer D, Allen F, Feine JS. The effectiveness of 2-implant overdentures - a pragmatic international multicentre study. J Oral Rehabil. 2011 Mar;38(3):176-84. doi: 10.1111/j.1365-2842.2010.02143.x. PMID 20704639
- [Background] Schimmel M, Christou P, Herrmann F, Muller F. A two-colour chewing gum test for masticatory efficiency: development of different assessment methods. J Oral Rehabil. 2007 Sep;34(9):671-8. doi: 10.1111/j.1365-2842.2007.01773.x. PMID 17716266
- [Background] Schimmel M, Christou P, Miyazaki H, Halazonetis D, Herrmann FR, Muller F. A novel colourimetric technique to assess chewing function using two-coloured specimens: Validation and application. J Dent. 2015 Aug;43(8):955-64. doi: 10.1016/j.jdent.2015.06.003. Epub 2015 Jun 22. PMID 26111925
- [Background] Sheiham A, Steele JG, Marcenes W, Lowe C, Finch S, Bates CJ, Prentice A, Walls AW. The relationship among dental status, nutrient intake, and nutritional status in older people. J Dent Res. 2001 Feb;80(2):408-13. doi: 10.1177/00220345010800020201. PMID 11332523
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Slotte C, Gronningsaeter A, Halmoy AM, Ohrnell LO, Mordenfeld A, Isaksson S, Johansson LA. Four-Millimeter-Long Posterior-Mandible Implants: 5-Year Outcomes of a Prospective Multicenter Study. Clin Implant Dent Relat Res. 2015 Oct;17 Suppl 2:e385-95. doi: 10.1111/cid.12252. Epub 2014 Jul 17. PMID 25041489
- [Background] Thomason JM, Feine J, Exley C, Moynihan P, Muller F, Naert I, Ellis JS, Barclay C, Butterworth C, Scott B, Lynch C, Stewardson D, Smith P, Welfare R, Hyde P, McAndrew R, Fenlon M, Barclay S, Barker D. Mandibular two implant-supported overdentures as the first choice standard of care for edentulous patients--the York Consensus Statement. Br Dent J. 2009 Aug 22;207(4):185-6. doi: 10.1038/sj.bdj.2009.728. PMID 19696851
- [Background] van der Bilt A. Assessment of mastication with implications for oral rehabilitation: a review. J Oral Rehabil. 2011 Oct;38(10):754-80. doi: 10.1111/j.1365-2842.2010.02197.x. Epub 2011 Jan 17. PMID 21241351
- [Background] van der Bilt A, Burgers M, van Kampen FM, Cune MS. Mandibular implant-supported overdentures and oral function. Clin Oral Implants Res. 2010 Nov;21(11):1209-13. doi: 10.1111/j.1600-0501.2010.01915.x. PMID 20572834
- [Background] van Kampen FM, van der Bilt A, Cune MS, Fontijn-Tekamp FA, Bosman F. Masticatory function with implant-supported overdentures. J Dent Res. 2004 Sep;83(9):708-11. doi: 10.1177/154405910408300910. PMID 15329377
- [Background] Woda A, Hennequin M, Peyron MA. Mastication in humans: finding a rationale. J Oral Rehabil. 2011 Oct;38(10):781-4. doi: 10.1111/j.1365-2842.2011.02235.x. No abstract available. PMID 22093138